CLINICAL TRIAL: NCT04650165
Title: 10-year Progression of Diabetic Retinopathy: Identification of Signs and Surrogate Outcomes
Acronym: PROGRESS10
Status: Completed | Type: Observational
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Responsible Party: Sponsor
Other Study IDs: CEC/011/20
Record Dates: First submitted 2020-11-25; First posted 2020-12-02 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To characterize both functionally and morphologically initial Diabetic Retinopathy (DR) stages and their progression over a period of 10 years.

DETAILED DESCRIPTION:
Diabetic retinopathy (DR) is the most frequent complication of diabetes mellitus and the leading cause of legal blindness in active populations of industrialized countries. Progression of DR has been up to now classified according to the ETDRS classification, based on a multicentric study that evaluated the effect of laser photocoagulation on advanced stages of DR. Although appropriate for late stages of DR, it does not grade progression well in the initial stages of the disease. Initial stages of DR require urgent characterization and their evolution should be well defined because some of the lesions are still reversible.

The early stages of DR are characterized by 4 main alterations: microaneurysms (MA) and retinal hemorrhages, represented by red dots in the fundus, blood-retinal barrier breakdown, capillary closure and damage of neuronal and glial cells of the retina. Thus, there are both microvascular changes, with endothelial cell and pericyte damage with thickening of basement membrane, and neuronal changes.

Based on previous studies, progression of DR does not occur at the same rate in all patients. Some never develop vision loss, whereas others rapidly progress to macular edema or neovascularization leading to vision loss. The understanding of the mechanisms that balance in different direction is of outmost importance. The duration of diabetes mellitus and the metabolic control are major risk factors for DR progression, but they are insufficient to explain the great variability observed in patients.

Recent data indicate that MA turnover may be an appropriate indicator of DR progression. Our research group has identified different DR progression phenotypes. Phenotype A is characterized by a low MA turnover, phenotype B characterized by increased thickness and phenotype C with predominant ischemia, with a high MA turnover. These phenotypes were defined based on MA turnover (RetmarkerDR) and on central retinal thickness (RT) measured by Optical Coherence Tomography (OCT) and the model was able to correctly identify eyes at risk of progression. 61,8-76,7% of eyes with an increase RT in the central subfield, inner and/or outer ring allowed a MA formation rate ≥ 2 and/or a MA turnover ≥ 6. More recently, some genetic variants have been linked to the different phenotypes and may explain specific progression patterns.

There is emerging evidence to suggest that retinal neurodegeneration is an early event in the pathogenesis of DR and that it could participate in the development of microvascular abnormalities. The understanding of the underlying mechanisms leading to neurodegeneration and the identification of the mediators between neurodegeneration and microangiopathy is essential.

The Investigators aim to understand the extent of these cell abnormalities in the initial stages of DR and to characterize their progression.

Analysis of retinal thickness using OCT offers non-invasive evaluation of retinal edema and can suggest an appropriate treatment target. The Investigators will use recent and innovative approaches as Spectral domain OCT (SD-OCT) with retinal layers segmentation to study neurodegenerative changes occurring in DR. OCT-Angiography and OCT-Leakage layer by layer analysis will be used for microvasculature and blood retinal barrier assessment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have participated in the PROGRESS study;
* Subjects capable of understanding the information about the study and to give their informed consent to enter the study.
* Subjects willing and able to comply with the study

Exclusion Criteria:

- Inadequate ocular media and/ or pupil dilatation that interfere with fundus examinations

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects older than 50 years-old with type 2 Diabetes mellitus and no Diabetic Retinopathy or mild Non-Proliferative Diabetic Retinopathy who have participated in the PROGRESS study (NCT03010397).
Sampling Method: Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Phenotypic classification of DR in a 5-year period | 5 years
  Presence CME (Central Macular Edema) or PDR (Proliferative Diabetic Retinopathy)
DR severity level | 5 years
  Early Treatment Diabetic Retinopathy Study Research Group, grading (7 fields-CFP)

SECONDARY OUTCOMES:
Choroidal thickness analysis | 5 years
  Choroidal thickness assessed by Enhanced Depth Imaging (EDI) SD-OCT
Retinal thickness analysis | 5 years
  Retinal thickness (RT) in central subfield, inner and outer rings, assessed by SD-OCT and using layer-by-layer segmentation
Ellipsoid zone analysis | 5 years
  Degree of integrity of the ellipsoid zone, assessed by SD-OCT
SD- OCT- Angiography analysis | 5 years
  Vessel analysis, assessed by SD-OCT OCT-Angiography
OCT-Leakage analysis | 5 years
  LOR (low optical reflectivity) ratio in central subfield, inner and outer ring for assessment of BRB breakdown, assessed by OCT-Leakage
Retinal thickness quantification | 5 years
  Retinal nerve fiber layer thickness (RNFL) and ganglion cells layer (GCL) + inner plexiform layer thickness (IPL) thickness, assessed by layer-by-layer SD-OCT
mfERG assessement | 5 years
  P1 implicit time and P1 amplitude by ring

CONTACTS AND LOCATIONS:
Overall Officials: Inês P Marques, MD, Principal Investigator — AIBILI - Association for Innovation and Biomedical Research on Light and Image
Locations (1):
- AIBILI - Association for Innovation and Biomedical Research on Light and Image, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: Undecided